CLINICAL TRIAL: NCT03503331
Title: UAB Alzheimer's Disease Center Core Cohort - Imaging Substudy
Acronym: PiB ADC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jonathan E McConathy, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300001005; 1P30AG086401-01 (NIH)
Record Dates: First submitted 2018-02-26; First posted 2018-04-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Brain amyloid PET levels will be measured with the PET tracer [C-11]PiB in all study participants.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [C-11]PiB-PET/MRI (Experimental): All participants in this study will undergo an amyloid-PET imaging using the tracer [C-11]PiB with a simultaneous PET/MRI system. The [C-11]PiB dosage is 300-670 MBq (8 - 18 mCi) given intravenously, and the PET/MRI imaging time is approximately 60 min.
  Interventions: Drug: [C-11]PiB-PET/MRI

INTERVENTIONS:
Drug: [C-11]PiB-PET/MRI — All study participants will undergo brain imaging with [C-11]PiB-PET/MRI. [C-11]PiB is a PET imaging agent used primarily to measure the amount of abnormal protein (called beta-amyloid) in the brain. The investigator will also use this tracer to evaluate regional cerebral blood flow.

SUMMARY:
The primary objective of this study is to measure the concentration and the regional brain distribution of pathologic amyloid deposition using the PET tracer [C-11]PiB in participants in the UAB Alzheimer's Disease Center cohort. Assessment of interactions between race and vascular risk factors, brain amyloid levels measured with [C-11]PiB-PET, and cognitive status will be the primary outcome of this imaging study.

DETAILED DESCRIPTION:
The primary objective of this study is to measure the concentration and the regional brain distribution of pathologic amyloid deposition using the PET tracer [C-11]PiB in participants in the UAB-ADC cohort. The amount and distribution of [C-11]PiB in the brain will be correlated to demographic, clinical, genetic, and biospecimen data acquired through the separate ongoing UAB-ADC study. Assessment of interactions between race and vascular risk factors, brain amyloid levels measured with [C-11]PiB-PET, and cognitive status will be the primary outcome of this imaging study. As a secondary aim, the investigators will assess the ability of the early flow frames from [C-11]PiB-PET and brain volumetric measurements with MRI to serve as a marker of neuronal injury and to predict cognitive status in conjunction with the amyloid-PET results.

ELIGIBILITY:
Inclusion Criteria:

- 1. Enrollment in the UAB-ADC study under a separate IRB-approved research protocol (IRB-300000169).

2. Negative urine or serum B-hCG test within 2 days of [C-11]PiB administration in women of child bearing potential. Women who are post-menopausal with at least 1 year since last menses or documented surgical sterilization will not require pregnancy testing.

Exclusion Criteria:

1. Meets any exclusion criteria for the UAB-ADC study (IRB-300000169).
2. Inability or contraindication for undergoing MRI and/or PET imaging
3. Inability to participate in the imaging studies due to severity of dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of pathological beta-amyloid in the brain | 5 years
  The amount of pathological beta-amyloid in the brains of study participants will be measured with [C-11]PiB-PET/MRI using standardized uptake value ratios (SUVRs) derived from the PET images.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States